CLINICAL TRIAL: NCT00657241
Title: Cardioprotective Benefits of Carvedilol-CR or Valsartan Added to Lisinopril
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, JOSEPH IZZO, Professor of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 111704
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Hypertension
Keywords: cardiac work; carvedilol CR; valsartan; tonometry
MeSH Terms: conditions — Hypertension | interventions — Carvedilol; Valsartan

STUDY DESIGN:
Intervention Model Description: Run-in period with lisinopril is followed by random entry into valsartan followed by carvedilol CR or carvedilol CR followed by valsartan
Who Masked: Participant
Masking Description: Drugs names omitted on patient bottles
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (A) ARB first, beta-blocker second (Active Comparator): Valsartan 160 mg daily (one week) and valsartan 320 mg daily (3 weeks) followed by carvedilol CR 20 mg daily (one week) and carvedilol CR 40 mg daily (3 weeks)
  Interventions: Drug: Carvedilol CR; Drug: Valsartan
- (B) Beta-blocker first, ARB second (Active Comparator): carvedilol CR 20 mg daily (one week) and carvedilol CR 40 mg daily (3 weeks) followed by valsartan 160 mg daily (1 week) and valsartan 320 mg daily (3 weeks).
  Interventions: Drug: Carvedilol CR; Drug: Valsartan

INTERVENTIONS:
Drug: Carvedilol CR
  Other Names: Coreg CR
Drug: Valsartan
  Other Names: Diovan

SUMMARY:
14-week single blind, double baseline, forced-titration, cross-over comparison of the cardiac benefits of Coreg CR compared to valsartan added to existing ACE inhibition

DETAILED DESCRIPTION:
Combination drug therapy is necessary for optimal blood pressure reduction and current guidelines mandate the concomitant use of ACE inhibitors and β-blockers in most patients at significant risk for cardiovascular disease (CVD) events. There is also continuing interest in combining angiotensin receptor blockers (ARBs) with ACE inhibitors in hypertension based on the unsubstantiated belief that "more complete" renin-angiotensin system inhibition is desirable. It is more attractive physiologically to combine a long-acting β-blocker with vasodilatory actions (carvedilol CR) with an ACE inhibitor because this combination addresses more directly the two fundamental hemodynamic changes needed to reduce CVD events: lowering systolic BP (afterload) and lowering heart rate; the product of the two is a reliable surrogate for reduced cardiac work. In fact, clinical trial data suggest that there is no appreciable additional BP lowering when ARBs are added to ACE inhibitors and neither class lowers heart rate. The present proposal is designed to demonstrate the superior "cardioprotection" of carvedilol CR compared to ARB (valsartan) when each is added to background ACE inhibitor therapy. Principal dependent variables include ambulatory cardiac work (24-hour mean ambulatory systolic BP x heart rate) and laboratory stress responses (central systolic time-tension indices derived from arterial tonometry pre- and post-bicycle exercise). Secondary hemodynamic variables will define changes in flow and pressure (e.g. central systolic BP and forward and reflected pressure wave estimations).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with residual (uncontrolled) hypertension on lisinopril monotherapy, defined as 24-hour ambulatory diastolic BP >85 mmHg.

Exclusion Criteria:

A subject meeting any of the following conditions will be excluded from the study:

* History of serious adverse effects with ACE inhibitor, Coreg, or valsartan
* Known or suspected causes of secondary hypertension (e.g., renovascular stenosis, primary hyperaldosteronism)
* Known ischemic heart disease requiring beta-blocker therapy (includes angina, prior transmural myocardial infarction, coronary artery bypass graft surgery or percutaneous transluminal coronary angioplasty or stenting within 6 months prior to study entry).
* Heart failure (NYHA Functional Class II-IV)
* Obstructive valvular heart disease or obstructive hypertrophic cardiomyopathy
* Presence of clinically significant ventricular or supraventricular arrhythmias (e.g. atrial fibrillation/flutter), pre-excitation syndrome, second or third degree AV block, other conduction defects necessitating the implantation of a permanent cardiac pacemaker, or sick sinus syndrome.
* Chronic kidney disease (serum creatinine >2.5 within past 6 months)
* Uncontrolled diabetes mellitus (i.e., a fasting blood glucose >200 mg/dL [>11.1 mmol/L] or hemoglobin A1c > 10%
* History of alcohol or other drug abuse within 6 months prior to enrollment
* Concomitant treatment or probable need for treatment with prohibited medications. NSAIDs, diabetes medications and other chronic meds are permitted if continued throughout study without dosage change.
* Any other medical condition which renders the subject unable to complete the study or which would interfere with optimal participation in the study or produce a significant risk to the subject
* Those with persistent systolic BP elevations above 179 mmHg will be discontinued from the study as will those with any significant adverse effect of medication.
* Positive pregnancy test or failure to practice adequate contraception in women of child-bearing potential
* Bronchospastic asthma requiring chronic steroid or inhaler therapy
* Any women with child-bearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Izzo, M.D., Principal Investigator — SUNY Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Izzo JL Jr, Yedlapati SH, Faheem SM, Younus U, Osmond PJ. Differences in mean and variability of heart rate and ambulatory rate-pressure product when valsartan or carvedilol is added to lisinopril. J Am Soc Hypertens. 2012 Nov-Dec;6(6):399-404. doi: 10.1016/j.jash.2012.08.007. Epub 2012 Oct 26. PMID 23107894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited by advertisement or from the practice of the PI
Pre-assignment Details: Prior antihypertensive medications were discontinued and subjects entered a 3-week run-in taking lisinopril 40 mg daily
Groups:
- ARB First: Lisinopril 40 mg daily plus valsartan 160 mg daily (one week) then valsartan 320 mg daily (3 weeks) followed by lisinopril 40 mg daily plus carvedilol CR 20 mg daily (one week) then carvedilol CR 40 mg daily (3 weeks)
- Beta-blocker First: Lisinopril 40 mg daily plus carvedilol CR 20 mg (one week) and carvedilol CR 40 mg (3 weeks) followed by lisinopril 40 mg daily plus valsartan 160 mg daily (one week) and valsartan 320 mg daily (3 weeks).
Period: Overall Study
Arm/Group | ARB First | Beta-blocker First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since all 30 participants will receive both drugs, the effects of the 2 drugs on the experimental endpoints will be compared by paired t-test. The 2 study arms refer to the randomization of sequential drug use (ARB first or beta-blocker first), which is designed to guard against the order (carryover) bias that might occur is the same drug sequence was used for all participants.
Groups:
- ARB First: Lisinopril 40 mg daily plus valsartan 160 mg daily (one week) then valsartan 320 mg daily (3 weeks) followed by lisinopril 40 mg daily plus carvedilol CR 20 mg daily (1 week) then carvedilol CR 40 mg daily (3 weeks)
- Beta-blocker First: Lisinopril 40 mg daily plus carvedilol CR 20 mg daily (1 week) then carvedilol CR 40 mg daily (3 weeks) followed by lisinopril 40 mg daily plus valsartan 160 mg daily (one week) then valsartan 320 mg daily (3 weeks)
- Total: Total of all reporting groups
Arm/Group | ARB First | Beta-blocker First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9.5) | 56 (9.5) | 56 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Difference in Resting CTTI Between Carvedilol CR (Beta-blocker) and Valsartan (ARB) in Combination With Lisinopril.
Description: Cardiac time-tension index (CTTI) is a refined version of the rate-pressure product (RPP, historically systolic [S] BP x heart rate) reported by the SphygmoCor pulse wave analysis system used in this trial. CTTI is preferable to RPP because the latter overestimates the contribution of systolic BP to cardiac work (the formula intrinsically assumes maximum SBP throughout the entire heart period [RR interval]). In contrast, CTTI represents cardiac work during the actual systolic time interval (STI, the period of active contraction, which is about 320 ms, inversely related to HR). Thus, CTTI = [mean systolic BP during STI, mmHg] x [STI/RR] x [HR, beats/min] and is expressed as "CTTI units" or as "mmHg*beats/min". Mean resting CTTI for SBP 150, HR 60 = about 2500 units (corresponding RPP = 9000 units). In this crossover study, the principal dependent variable is the mean within-subjects difference in supine CTTI between valsartan and carvedilol CR after 4 weeks of each treatment.
Time Frame: End of each treatment period (4 weeks on ARB or beta-blocker)
Population: Analysis groups are different from treatment arms, which reflect the sequence of administration of the comparators, valsartan or carvedilol CR, which are received by all participants. CTTI comparisons made at end of each 4-week treatment period; study powered to detect an 8% difference in CTTI by paired t-test at p < 0.05, power 0.8.
Measure: Mean (Standard Deviation); unit: CTTI units (mmHg*beats/min)
Groups:
- Carvedilol CR: Lisinopril 40 mg daily plus carvedilol CR 20 mg (one week) then carvedilol CR 40 mg (3 weeks) administered first or second
- Valsartan: lisinopril 40 mg daily plus valsartan 160 mg daily (1 week) then valsartan 320 mg daily (3 weeks) administered first or second
Arm/Group | Carvedilol CR | Valsartan
Number analyzed (Participants) | 30 | 30
CTTI units (mmHg*beats/min) | 2447 (547) | 2500 (561)
Statistical Analysis 1: Comparison: Carvedilol CR vs Valsartan; Statistical analysis performed on treatment groups (valsartan or carvedilol CR) at end of treatment period (4 weeks), not on the randomization arms in the crossover design (which controlled for carryover effects of the prior treatment arm); Test type: Superiority — All hemodynamic variables are continuous and all participants received both treatments, so paired-t analysis could be used. While paired t-tests do not necessarily require a power and sample size analysis, we estimated that 30 subjects were sufficient to detect an 8% difference in CTTI between comparators at p<0.05 with a conservatively estimated power of 0.8; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Heart Rate (Beats/Min)
Description: Hemodynamic variable (cardiac rate)
Time Frame: End of each treatment period (4 weeks on ARB or beta-blocker)
Population: These analysis groups reflect the main study aim of direct comparison of ARB to beta-blocker with respect to cardiac work (CTTI). The analysis groups are not the same as the cross-over arms that represent sequence of drug administration (i.e. "ARB first" or "beta-blocker first").
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Lisinopril Plus Valsartan: Lisinopril 40 mg daily plus valsartan 160 mg daily (one week) followed by lisinopril 40 mg daily plus valsartan 320 mg (3 weeks)
- Lisinopril Plus Carvedilol: Lisinopril 40 mg daily plus carvedilol CR 20 mg (one week) followed by lisinopril 40 mg daily plus carvedilol CR 40 mg (3 weeks).
Arm/Group | Lisinopril Plus Valsartan | Lisinopril Plus Carvedilol
Number analyzed (Participants) | 30 | 30
beats per minute | 75 (17) | 68 (14)

3. Secondary Outcome: Stroke Volume (SV)
Description: Hemodynamic variable (volume pumped per heart beat) in mL per beat. Clinically, SV is reported simply as mL
Time Frame: End of each treatment period (4 weeks on ARB or beta-blocker)
Population: Mean of (intra-individual) SV values after 4 weeks of valsartan or carvedilol CR
Measure: Mean (Standard Deviation); unit: mL or mL/beat
Arm/Group | Lisinopril Plus Valsartan | Lisinopril Plus Carvedilol
Number analyzed (Participants) | 30 | 30
mL or mL/beat | 77 (17) | 76 (15)
Statistical Analysis 1: Comparison: Lisinopril Plus Valsartan vs Lisinopril Plus Carvedilol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, t-test, 2 sided; paired t-test

4. Secondary Outcome: Cardiac Output
Description: Hemodynamic variable representing whole-body blood flow (the product of heart rate and stroke volume)
Time Frame: End of each 4-week treatment period (valsartan vs. carvedilol CR)
Population: 4-week treatment period (valsartan vs. carvedilol CR); comparison by paired t-test
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Lisinopril Plus Valsartan: Lisinopril 40 mg daily plus valsartan 160 mg daily (one week)followed by lisinopril 40 mg daily plus valsartan 320 mg (3 weeks)
- Lisinopril Plus Carvedilol: Lisinopril 40 mg daily plus Coreg CR 20 mg (one week) followed by lisinopril 40 mg daily plus Coreg CR 40 mg (3 weeks).
Arm/Group | Lisinopril Plus Valsartan | Lisinopril Plus Carvedilol
Number analyzed (Participants) | 30 | 30
L/min | 5.7 (1.4) | 5.1 (1.1)
Statistical Analysis 1: Comparison: Lisinopril Plus Valsartan vs Lisinopril Plus Carvedilol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, t-test, 2 sided; Paired t-test

5. Secondary Outcome: Systemic Vascular Resistance
Description: Hemodynamic variable measured as mean arterial pressure (mmHg) / cardiac output (L/min) *80 in units of dyne-sec-cm[-5]
Time Frame: End of each treatment period (4 weeks of valsartan or carvedilol CR)
Population: Valsartan vs. carvedilol CR at end of 4-week treatment period; comparison by paired t-test
Measure: Mean (Standard Deviation); unit: dyne sec cm-5
Arm/Group | Lisinopril Plus Valsartan | Lisinopril Plus Carvedilol
Number analyzed (Participants) | 30 | 30
dyne sec cm-5 | 1407 (378) | 1591 (410)
Statistical Analysis 1: Comparison: Lisinopril Plus Valsartan vs Lisinopril Plus Carvedilol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, t-test, 2 sided; paired t-test

6. Secondary Outcome: Central Systolic Blood Pressure
Description: Aortic SBP derived non-invasively from radial arterial tonometry, pulse wave analysis, and a generalized transfer function algorithm within the SphygmoCor device. Aortic SBP is different from brachial SBP and is variably lower than brachial SBP due to pulse wave transmission differences between individuals. It is expressed in mmHg.
Time Frame: End of each treatment period (4 weeks of valsartan or carvedilol CR)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril Plus Valsartan | Lisinopril Plus Carvedilol
Number analyzed (Participants) | 30 | 30
mmHg | 130 (22) | 141 (25)
Statistical Analysis 1: Comparison: Lisinopril Plus Valsartan vs Lisinopril Plus Carvedilol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, t-test, 2 sided; paired t-test

ADVERSE EVENTS:
Time Frame: 9 weeks (duration of the crossover study, including 4 weeks each of valsartan or carvedilol in random order and 1 week of follow-up)
Description: Standard definitions
Groups:
- Valsartan: Lisinopril 40 mg daily plus valsartan 160 mg daily (one week) then valsartan 320 mg daily (3 weeks)
- Carvedilol CR: Lisinopril 40 mg daily plus carvedilol CR 20 mg daily (one week) then carvedilol CR 40 mg daily (3 weeks).
Arm/Group | Valsartan | Carvedilol CR
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Short duration of trial may miss long-term effects. Statistical powering for primary outcome may preclude secondary analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No